CLINICAL TRIAL: NCT02724891
Title: Validation of Electronic (Web-based and Smartphone) Administration of Measures of Pelvic Floor Dysfunction
Brief Title: Web-based Validation Pelvic Floor Questionnaires
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of Wisconsin, Madison (Other); University of Arkansas (Other); The Methodist Hospital Research Institute (Other); University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: AAAO8451
Record Dates: First submitted 2016-02-04; First posted 2016-03-31 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Pelvic Floor Dysfunction
Keywords: Pelvic Floor Dysfunction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1 paper form first: paper questionnaires first then web/smart phone questionnaires after a 2-week washout period
  Interventions: Other: paper form; Other: web/smartphone form
- Arm 2 web/smartphone form first: web/smart phone questionnaires first then paper questionnaires after a 2-week washout period
  Interventions: Other: paper form; Other: web/smartphone form

INTERVENTIONS:
Other: paper form — questionnaires in paper form
Other: web/smartphone form — questionnaires in web/smartphone

SUMMARY:
Patient-reported outcomes are commonly used in healthcare. Examples include validated symptom-based questionnaires and health diaries. In the field of Female Pelvic Medicine and Reconstructive Surgery there are many questionnaires and diaries that have been validated for a paper-based administration. As technology is incorporated into delivery of medical care and research, investigators need to consider how to collect data electronically while ensuring that this new format is equivalent to the paper questionnaires they rely on. In this study, the investigators aim to validate a series of validated questionnaires and symptom diaries administered via the web and smartphone for a more streamlined care for the patients.

DETAILED DESCRIPTION:
Health questionnaires and health diaries are two forms of patient-reported outcomes (PRO) commonly used in healthcare. Health questionnaires are often used as intake logs, discerning and recording the symptoms and severity of a problem at the time of presentation. Health diaries, in contrast, are ongoing logs which allow for mindful attention to symptoms and monitoring of response to therapy. Unfortunately, both types of PRO forms are often under-utilized or uninterpretable because they are collected on paper. Within urogynecology, PRO scales such as the Pelvic Floor Distress Inventory (PFDI), Pelvic Floor Impact Questionnaire (PFIQ), Bristol Stool Chart, Bladder Diaries and others are used ubiquitously. Their impact, however, is diminished by poor compliance and recall bias. The move towards electronic PRO measures would be endorsed by patients (who can track and interact with their data), physicians (who can track progress and study group outcomes) and by regulators (who want to ensure accurate and reproducible data collection). Electronic PRO tools, particularly on the patient's own device, would allow for increased rate of reporting through mobile availability, time stamping of data to prevent recall bias and reduction in data entry mistakes and costs.

Study Procedures After informed consent is obtained, demographic data will be collected. Subjects will be administered the questionnaires either in paper or web-based or smartphone form based on a random number block scheme. At least two weeks later but prior to treatment they will complete the other form of the questionnaire. This can occur at their next office visit or can be completed at home. Subjects will be emailed and/or called by research staff to remind them to complete the second set of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age presenting with pelvic floor dysfunction

Exclusion Criteria:

* Unable to repeat questionnaires or return to the office in 2 weeks
* No access to computer/web or smartphone
* Pregnancy (as gestational age will advance during 2 week time interval and symptoms may change)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective validation study. Subjects will be recruited at their visit to the Female Pelvic Medicine and Reconstructive Surgery offices and clinics at Columbia and Cornell. Demographic information will be collected at the initial visit/enrollment including age, race, parity, and presenting complaint.
  Questionnaires will be administered based on a randomization scheme. These include:
  * Pelvic Floor Disorders Inventory short form (PFDI-20)
  * Pelvic Floor Impact Questionnaire (PFIQ-7)
  * Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)
  * Bristol Stool Scale (BSS)
  Questionnaires will be administered via paper-based form, web-based, or smartphone app based on randomization scheme.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Test-retest reliability of PFDI-20 in the electronic format | minimum 2 week interval until subject receives treatment for the condition or up to one year
  Subjects will complete the paper and either web-based or smartphone versions of the PFDI-20 with at least a 2 week interval between administration of the 2 versions.
Test-retest reliability of PFIQ-7 in the electronic format | minimum 2 week interval until subject receives treatment for the condition or up to one year
  Subjects will complete the paper and either web-based or smartphone versions of the PFIQ-7 with at least a 2 week interval between administration of the 2 versions.
Test-retest reliability of PISQ-12 in the electronic format | minimum 2 week interval until subject receives treatment for the condition or up to one year
  Subjects will complete the paper and either web-based or smartphone versions of the PISQ-12 with at least a 2 week interval between administration of the 2 versions.
Test-retest reliability of BSS in the electronic format | minimum 2 week interval until subject receives treatment for the condition or up to one year
  Subjects will complete the paper and either web-based or smartphone versions of the BSS with at least a 2 week interval between administration of the 2 versions.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Grimes, MD, Principal Investigator — Columbia University
Locations (5):
- United States (4):
  - University of Arkansas, Fayetteville, Arkansas
  - Columbia University Irving Medical Center, New York, New York
  - Houston Methodist Hospital, Houston, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimes CL, Antosh DD, Oliphant S, Yurteri-Kaplan L, Kim-Fine S, Melamud G, Heisler C, Chung DE; Collaborative Research in Pelvic Surgery Consortium (CoRPS). Correlation of Electronic (Web-Based and Smartphone) Administration of Measures of Pelvic Floor Dysfunction: A Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2020 Jun;26(6):396-400. doi: 10.1097/SPV.0000000000000713. PMID 30889034